CLINICAL TRIAL: NCT03332589
Title: A Phase 1 Study of E6201 Plus Dabrafenib for the Treatment of Central Nervous System Metastases (CNS) From BRAF V600-Mutated Metastatic Melanoma
Brief Title: E6201 Plus Dabrafenib for the Treatment of Metastatic Melanoma Central Nervous System Metastases (CNS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Single center study: Principal Investigator left institution.
Sponsor: Spirita Oncology, LLC (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STX-101-02
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-12

CONDITIONS: Malignant Melanoma; Brain Metastases
Keywords: Melanoma; CNS metastases; BRAF V600 mutation; E6201; Dabrafenib
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — 14-(ethylamino)-8,9,16-trihydroxy-3,4-dimethyl-3,4,9,19-tetrahydro-1H-2-benzoxacyclotetradecine-1,7(8H)-dione; dabrafenib

STUDY DESIGN:
Intervention Model Description: 4 subjects were treated in the E6201 Monotherapy Safety Run-in Phase. A total of 6-12 subjects are anticipated in the E6201 plus dabrafenib Combination Safety Run-in Phase. Once an MTD of the combination is determined, a total of 6 subjects will be treated at the combined MTD before the Expansion Phase will begin. In the Expansion Phase, an additional cohort of up to N=18 subjects will be treated at the combined E6201 plus dabrafenib MTD. Subjects treated at the MTD in the Combination Safety Run-in Phase will count towards accrual in the Expansion Phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy Safety Run-in: E6201 (Experimental): E6201 320 mg/m^2 administered IV over 2 hours twice weekly on Days 1, 4, 8, 11, 15 and 18, repeated every 28 days (=1 cycle).
  Dose reductions for toxicity are 240 mg/m^2 (Dose Level -1) and 160 mg/m^2 (Dose Level -2) twice weekly.
  Interventions: Drug: E6201
- Combination Safety Run-in: E6201 Plus Dabrafenib (Experimental): Dose Level 1: E6201 320 mg/m^2 twice weekly plus dabrafenib 150 mg BID. Dose Level -1: E6201 240 mg/m^2 twice weekly plus dabrafenib 150 mg BID. Dose Level -2: E6201 240 mg/m^2 twice weekly plus dabrafenib 100 mg BID. Dose Level -3: E6201 160 mg/m^2 twice weekly plus dabrafenib 100 mg BID Dose Level -4: E6201 160 mg/m^2 twice weekly plus dabrafenib 75 mg BID. Dose Level -5: E6201 160 mg/m^2 twice weekly plus dabrafenib 50 mg BID.
  Interventions: Drug: E6201 plus dabrafenib
- Expansion: E6201 Plus Dabrafenib (Experimental): A total of up to N=18 will be treated at the E6201 plus dabrafenib combined MTD.
  Interventions: Drug: E6201 plus dabrafenib

INTERVENTIONS:
Drug: E6201 — E6201 formulated in cyclodextrin for IV administration.
  Arms: Monotherapy Safety Run-in: E6201
Drug: E6201 plus dabrafenib — E6201 formulated in cyclodextrin for IV administration. Dabrafenib capsules for oral administration.
  Arms: Combination Safety Run-in: E6201 Plus Dabrafenib; Expansion: E6201 Plus Dabrafenib

SUMMARY:
This is a Phase 1 study of E6201 plus dabrafenib for the treatment of CNS metastases in BRAF V600-mutated metastatic melanoma. A total of up to N=28-34 subjects with melanoma metastasized to the CNS will be included.

DETAILED DESCRIPTION:
Selected subjects will be: both males and females age ≥18 years; histologically confirmed melanoma with BRAF V600 mutation with CNS metastasis; archived tumor sample from the primary, recurrent or metastatic disease with documented BRAF mutation; recovered from all acute toxicities (≤ Grade 1) due to prior immunotherapy; determined to have adequate renal and hepatic function, and no known history of significant cardiac disease.

Monotherapy Safety Run-in Phase: Following screening, a total of up to 4 subjects were enrolled. E6201 was administered by intravenous (IV) infusion over a 2-hour period at a dose of 320 mg/m^2 twice weekly (Days 1, 4, 8, 11, 15 and 18) for three weeks, repeated every 28 days (1 cycle) until progression of disease, observation of unacceptable adverse events, intercurrent illness or changes in the subject's condition that prevents further study participation.

Combination Safety Run-in Phase: Following screening, a total of 6-12 subjects are anticipated to establish the recommended doses of E6201 plus dabrafenib. E6201 will be administered by IV infusion over a 2-hour period twice weekly (Days 1, 4, 8, 11, 15 and 18) repeated every 28 days plus dabrafenib orally twice daily (=1 cycle).

Dose Level 1: E6201 320 mg/m^2 twice weekly plus dabrafenib 150 mg BID. Dose Level -1: E6201 240 mg/m^2 twice weekly plus dabrafenib 150 mg BID. Dose Level -2: E6201 240 mg/m^2 twice weekly plus dabrafenib 100 mg BID. Dose Level -3: E6201 160 mg/m^2 twice weekly plus dabrafenib 100 mg BID Dose Level -4: E6201 160 mg/m^2 twice weekly plus dabrafenib 75 mg BID. Dose Level -5: E6201 160 mg/m^2 twice weekly plus dabrafenib 50 mg BID.

A total of 6 subjects will be treated at the combined MTD doses for both drugs in the Combination Safety Run-in Phase before beginning the Expansion Phase.

Expansion Phase: An additional cohort of up to N=18 subjects will be treated at the E6201 plus dabrafenib combined MTD. Subjects treated at the MTD in the Combination Safety Run-in Phase will count towards accrual in the Expansion Phase.

CNS disease response will be assessed according to 2 methodologies: Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1) and Response Assessment in Neuro-Oncology - Brain Metastases (RANO-BM). Non-CNS systemic disease will be assessed according to RECIST v. 1.1.

Blood for hematology and serum chemistry determinations will be collected and ECGs will be taken during the study. Assessments will be obtained at Week 8 and every 8 weeks thereafter until documented progression of disease (PD). Subjects who demonstrate clinical benefit will be allowed to continue therapy with E6201 until progression of disease, observation of unacceptable adverse events, intercurrent illness or changes in the subject's condition that prevents further study participation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Histologically or cytologically confirmed BRAFV600-mutated melanoma
* Documented metastasis of the primary tumor to the CNS
* BRAF-mutation melanoma tumor status will be established prior to entry based on previous BRAF-gene analysis or MEK pathway mutation reports from a CLIA qualified laboratory. If a report is not available, the mutation analysis will be performed at Screening on archival tissue
* Other metastatic melanoma systemic disease allowed
* At least one measurable brain metastasis, 0.5 - 3.0 cm, as assessed by MRI ≤ 3 weeks prior to initiation of study treatment, provided neurological sequelae have resolved completely and at least one measurable metastasis with documented disease progression is present on MRI
* Prior stereotactic radiosurgery and/or excision of up to 3 brain metastases is allowed > 3 weeks before initiation of study treatment, provided neurological sequelae have resolved completely and at least one measurable metastasis with documented disease progression is present on MRI
* One prior line of immunotherapy for metastatic disease is allowed, if ≥ 2 weeks has elapsed between the end of therapy and initiation of study treatment
* Prior melanoma adjuvant immunotherapy is allowed, if ≥ 6 months has elapsed between the end of therapy and initiation of study treatment
* Prior melanoma adjuvant BRAF/MEK inhibitor therapy is allowed, if ≥ 12 months has elapsed between the end of therapy and initiation of study treatment
* Able to swallow and retain oral medication with no clinically significant gastrointestinal abnormalities that may alter absorption, such as malabsorption syndrome or major resection of the stomach or bowels (Combination Safety Run-in and Expansion Phases of the study only)
* Asymptomatic or symptomatic CNS metastasis is allowed
* Stable dose of corticosteroids for CNS metastasis for ≥ 7 days allowed
* Patients with seizures due to CNS metastases must be controlled with stable anti-epileptic treatment for ≥ 14 days
* Bisphosphonates and/or denosumab are allowed
* Adequate performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy of ≥ 3 months
* Adequate hematologic parameters without ongoing transfusional support:

  * Hemoglobin (Hb) ≥ 9 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9 cells/L
  * Platelets ≥ 75 x 10^9 cells/L
* Adequate renal and hepatic function:

  * Creatinine ≤ 1.5 x the upper limit of normal (ULN), or calculated creatinine clearance ≥ 50 mL/minute x 1.73 m^2
  * Total bilirubin ≤ 2 times the upper limit of normal (ULN) unless due to Gilbert's disease
  * ALT/AST ≤ 2.5 times ULN, or < 5 times ULN for subjects with liver metastases
* Negative serum pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential (WCBP). Sexually active WCBP and male subjects must agree to use adequate methods to avoid pregnancy throughout the study and for 28 days after the completion of study treatment.
* Ability to provide written informed consent

Exclusion Criteria:

* Urgent need of treatment to prevent acute neurologic deterioration, including urgent neurosurgery or radiotherapy
* Symptoms of uncontrolled intracranial pressure
* Symptomatic or untreated spinal cord compression
* Prior treatment with any chemotherapeutic or investigational agent
* Prior treatment with any BRAF and/or MEK inhibitor for metastatic disease
* Prior treatment with > 1 line of immunotherapy for metastatic disease
* Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV
* QT interval corrected for rate (QTc) > 480 msec for on the ECG obtained at Screening using Fridericia method for QTc calculation
* Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) requiring systemic antiviral treatment within the last week prior to study treatment
* Other active infection requiring IV antibiotic usage within the last week prior to study treatment
* Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hani M Babiker, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated before any participants were enrolled in the Combination or Expansion Phases.
Groups:
- Monotherapy Safety Run-in: E6201: E6201 320 mg/m^2 administered IV over 2 hours twice weekly on Days 1, 4, 8, 11, 15 and 18, repeated every 28 days (=1 cycle).
  Dose reductions for toxicity are 240 mg/m^2 (Dose Level -1) and 160 mg/m^2 (Dose Level -2) twice weekly.
  E6201: E6201 for Injection formulated in cyclodextrin for IV administration
- Combination Safety Run-in: E6201 Plus Dabrafenib: Dose Level 1: E6201 320 mg/m^2 twice weekly plus dabrafenib 150 mg BID. Dose Level -1: E6201 240 mg/m^2 twice weekly plus dabrafenib 150 mg BID. Dose Level -2: E6201 240 mg/m^2 twice weekly plus dabrafenib 100 mg BID. Dose Level -3: E6201 160 mg/m^2 twice weekly plus dabrafenib 100 mg BID Dose Level -4: E6201 160 mg/m^2 twice weekly plus dabrafenib 75 mg BID. Dose Level -5: E6201 160 mg/m^2 twice weekly plus dabrafenib 50 mg BID.
  E6201 plus dabrafenib: E6201 for Injection formulated in cyclodextrin for IV administration plus oral dabrafenib capsules
- Expansion: E6201 Plus Dabrafenib: A total of up to N=18 will be treated at the E6201 plus dabrafenib combined MTD.
  E6201 plus dabrafenib: E6201 for Injection formulated in cyclodextrin for IV administration plus oral dabrafenib capsules
Period: Overall Study
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib
Started | 4 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in the Combination Safety Run-In or Expansion Phases of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib | Total
Number analyzed (Participants) | 4 | 0 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14.7) |  |  | 51 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  | 2
  Male | 2 |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 1
  Not Hispanic or Latino | 3 |  |  | 3
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 4 |  |  | 4
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 |  |  | 4
Eastern Cooperative Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status:
  0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
     = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  2. = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  Participants
    0 | 1 |  |  | 1
    1 | 2 |  |  | 2
    2 | 1 |  |  | 1
Prior Cancer Therapies [Median (Full Range); unit: regimens] | 5.5 [4 to 7] |  |  | 5.5 [4 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Disease Overall Response Rate by RANO-BM
Description: CNS disease response will be assessed by Response Assessment in Neuro-Oncology - Brain Metastases (RANO-BM)
Time Frame: At the end of Cycle 2 and every 2 cycles through 6 months following last dose of study drug (each cycle is 28 days) up to 1 year.
Population: The analysis population was the per-protocol set (PPS). The PPS included all participants in the full analysis set (FAS) who had a valid baseline and one or more post-treatment assessments for a specific measure. No participants were enrolled in the Combination Safety Run-In or Expansion Phases of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib
Number analyzed (Participants) | 4 | 0 | 0
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 2 | 0 | 0
  Progressive Disease | 1 | 0 | 0
  Not Evaluable | 1 | 0 | 0

2. Primary Outcome: Intracranial Disease Overall Response Rate by RECIST 1.1
Description: CNS disease response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib
Number analyzed (Participants) | 4 | 0 | 0
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 2 | 0 | 0
  Progressive Disease | 1 | 0 | 0
  Not Evaluable | 1 | 0 | 0

3. Secondary Outcome: Intracranial Disease Duration of Response
Description: Length of time from the first evidence of Objective Response (complete response or partial response) to the first evidence of progression
Time Frame: as for outcome 1
Population: There were no Objective Responses during the study. Thus, Duration of Response could not be calculated.
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Systemic Disease Overall Response Rate (Other Than in the CNS)
Description: Systemic disease response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1RECIST 1.1.
Time Frame: as for outcome 1
Population: The analysis population was the per-protocol set (PPS). The PPS included all participants in the full analysis set (FAS) who had a valid baseline and one or more post-treatment assessments for a specific measure. No subjects were enrolled in the Combination Safety Run-In or Expansion Phases of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib
Number analyzed (Participants) | 4 | 0 | 0
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 3 | 0 | 0
  Progressive Disease | 0 | 0 | 0
  Not Evaluable | 1 | 0 | 0

5. Secondary Outcome: Progression-Free Survival
Description: Length of time from the date of first administration of study drug to the first evidence of disease progression or death, whichever is earlier
Time Frame: From Cycle 1 Day 1 through 6 months following the last dose of study drug (each cycle is 28 days) up to 1 year.
Population: as for outcome 4
Measure: Median (Standard Deviation); unit: months
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib
Number analyzed (Participants) | 1 | 0 | 0
months | NA — NA: Median could not be estimated due to insufficient number of participants with the event. |  |

6. Secondary Outcome: Overall Survival
Description: Length of time from the date of first administration of study drug to the date of death from any cause
Time Frame: From Cycle 1 Day 1 through 6 months following the last dose of study drug or death, whichever is earlier (each cycle is 28 days) up to 1 year.
Population: as for outcome 4
Measure: Median (Standard Deviation); unit: months
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib
Number analyzed (Participants) | 1 | 0 | 0
months | NA — NA: Median could not be estimated due to insufficient number of participants with the event. |  |

ADVERSE EVENTS:
Time Frame: Adverse event data and all-cause mortality data were collected for each subject from C1D1 to 6 months after the last dose of study drug up to 1 year.
Description: Adverse events were reported for all study participants who were administered at least one dose of study medication.
Arm/Group | Monotherapy Safety Run-in: E6201 | Combination Safety Run-in: E6201 Plus Dabrafenib | Expansion: E6201 Plus Dabrafenib
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monotherapy Safety Run-in: E6201 (N=4) | Combination Safety Run-in: E6201 Plus Dabrafenib (N=0) | Expansion: E6201 Plus Dabrafenib (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monotherapy Safety Run-in: E6201 (N=4) | Combination Safety Run-in: E6201 Plus Dabrafenib (N=0) | Expansion: E6201 Plus Dabrafenib (N=0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the departure of the study PI from the institution, the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT03332589/Prot_SAP_000.pdf